CLINICAL TRIAL: NCT06098586
Title: Partial Wrist Denervation Versus Self-managed Exercise Therapy in Patients with Wrist Osteoarthritis: a Randomized Controlled Multicenter Trial
Brief Title: Wrist Denervation Vs Exercise in Wrist Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Elin Swärd, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-04885-01
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis Wrist

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data assessors and analysts will be masked for treatment allocation (covered wrist / anonymous data sheet).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-managed exercise therapy program (Active Comparator): Exercise program focusing on functional re-learning and strengthening of the musculoskeletal system with the aim to create a stable wrist that can be used in a pain-free manner in activities of daily living.
  Interventions: Behavioral: Self-managed exercise therapy program
- Partial wrist denervation (Active Comparator): AIN and PIN neurectomy through a dorsal approach as described by Berger (Berger, 1998).
  Interventions: Procedure: Partial wrist denervation

INTERVENTIONS:
Behavioral: Self-managed exercise therapy program — Exercise program focusing on functional re-learning and strengthening of the musculoskeletal system with the aim to create a stable wrist that can be used in a pain-free manner in activities of daily living.
  Arms: Self-managed exercise therapy program
Procedure: Partial wrist denervation — AIN and PIN neurectomy through a dorsal approach as described by Berger (Berger, 1998).
  Arms: Partial wrist denervation

SUMMARY:
A randomized controlled trial comparing partial wrist denervation to a self-managed exercise therapy program in 140 patients with wrist osteoarthritis.

DETAILED DESCRIPTION:
Backgroud:

High quality evidence regarding the effectiveness of non-operative and operative treatments in wrist osteoarthritis are lacking.

Aim:

To analyze:

1. Does partial wrist denervation and self-managed exercise therapy improve patient-reported outcomes, pain, grip strength and range of motion (ROM) in wrist OA?
2. Is any of the two treatment concepts partial wrist denervation and self-managed exercise therapy more efficient than the other in terms of patient-reported outcomes, pain relief, grip strength and range of motion?

Method:

A multicenter parallel group, two-arm, randomized, controlled, assessor blinded, trial of 140 patients. The study is conducted at the departments of hand surgery at Södersjukhuset Stockholm and Malmö University hospital.

Group1:

Self-managed exercise therapy program containing:

* Patient education:
* Exercise therapy program:

The exercise therapy program is designed by Sara Larsson (physiotherapist at the Department of hand surgery in Malmö, Sweden), influenced by previous studies on wrist stability and proprioception. Focus is on functional re-learning and strengthening of the musculoskeletal system with the aim to create a stable wrist that can be used in a pain-free manner in activities of daily living. The program consists of neuromuscular exercises that focus on coordination, wrist stability and strength.

Group 2:

Surgery will be performed under local anesthesia (+ blood-less field or wide-awake local anesthesia no torniquet (WALANT) according to the surgeon's preference) through a single dorsal incision. AIN and PIN neurectomy will be performed as described by Berger (Berger, 1998).

Primary outcome:

Patient Rated Wrist Evaluation (PRWE) score (0-100) (MacDermid et al., 1998) 12 months after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Chronic wrist pain (≥6 months) due to Scapholunate advanced collapse (SLAC) / Scaphoid non-union advanced collapse (SNAC) grade 1-3 osteoarthritis.
* Radiological signs of osteoarthritis on posteroanterior and lateral radiograph.

Exclusion Criteria:

* Previous PIN or AIN neurectomy.
* Rheumatoid arthritis or other chronic inflammatory arthritis.
* Symptomatic osteoarthritis in the distal radio-ulnar (DRU), Scapho-trapezio-trapezoid (STT) or thumb carpometacarpal (CMC) joints.
* Ongoing infection.
* Inability to co-operate with the follow-up protocol.
* Systemic or intra-articular glucocorticoids or intraarticular PRP or Hyaluronic acid injections in the affected joint within 3 months prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2027-11-15 (Estimated)

PRIMARY OUTCOMES:
PRWE | 6 months
  Patient Rated Wrist Evaluation (PRWE) score (0-100 (high score worse outcome)) (MacDermid et al., 1998)

SECONDARY OUTCOMES:
PRWE | 3 months
  Patient Rated Wrist Evaluation (PRWE) score (0-100 (high score worse outcome)) (MacDermid et al., 1998)
PRWE | 12 months
  Patient Rated Wrist Evaluation (PRWE) score (0-100 (high score worse outcome)) (MacDermid et al., 1998)
PRWE | 5 years
  Patient Rated Wrist Evaluation (PRWE) score (0-100 (high score worse outcome)) (MacDermid et al., 1998)
Pain NRS | 3 months
  Pain at rest and on load measured by a Numerical Rating Scale (NRS, 0-100 (higher score worse outcome) (Salaffi et al 2004)
Pain NRS | 6 months
  Pain at rest and on load measured by a Numerical Rating Scale (NRS, 0-100 (higher score worse outcome) (Salaffi et al 2004)
Pain NRS | 12 months
  Pain at rest and on load measured by a Numerical Rating Scale (NRS, 0-100 (higher score worse outcome) (Salaffi et al 2004)
Pain NRS | 5 years
  Pain at rest and on load measured by a Numerical Rating Scale (NRS, 0-100 (higher score worse outcome) (Salaffi et al 2004)
EQ5D | 3 months
  EQ-5D-5L (0-1 (higher score better outcome)) (Brooks, 1996)
EQ5D | 6 months
  EQ-5D-5L (0-1 (higher score better outcome)) (Brooks, 1996)
EQ5D | 12 months
  EQ-5D-5L (0-1 (higher score better outcome)) (Brooks, 1996)
EQ5D | 5 years
  EQ-5D-5L (0-1 (higher score better outcome)) (Brooks, 1996)
GROC | 3 months
  Global rating of change (GROC, -5-+5, higher score better outcome)
GROC | 6 months
  Global rating of change (GROC, -5-+5, higher score better outcome)
GROC | 12 months
  Global rating of change (GROC, -5-+5, higher score better outcome)
GROC | 5 years
  Global rating of change (GROC, -5-+5, higher score better outcome)
Pain catastrophizing | 3 months
  PCS (Pain catastrophizing scale, 0-52, higher score worse outcome) (Sullivan et al, 1995)
Pain catastrophizing | 6 months
  PCS (Pain catastrophizing scale, 0-52, higher score worse outcome) (Sullivan et al, 1995)
Pain catastrophizing | 12 months
  PCS (Pain catastrophizing scale, 0-52, higher score worse outcome) (Sullivan et al, 1995)
Pain catastrophizing | 5 years
  PCS (Pain catastrophizing scale, 0-52, higher score worse outcome) (Sullivan et al, 1995)
ROM | 3 months
  Range of motion (ROM) of the wrist.
ROM | 6 months
  Range of motion (ROM) of the wrist.
ROM | 12 months
  Range of motion (ROM) of the wrist.
ROM | 5 years
  Range of motion (ROM) of the wrist.
Grip | 3 months
  Grip strength (Jamar).
Grip | 6 months
  Grip strength (Jamar).
Grip | 12 months
  Grip strength (Jamar).
Grip | 5 years
  Grip strength (Jamar).
Complications | 3 months
  Complications related to treatment
Complications | 6 months
  Complications related to treatment
Complications | 12 months
  Complications related to treatment
Complications | 5 years
  Complications related to treatment
Radiology | 5 years
  Radiological grade of osteoarthritis 5 years after inclusion compared to baseline.
Cost | 12 months
  Differences in direct costs associated with treatment and indirect costs.
sick leave | 12 months
  length of sick leave
work | 12 months
  ability to return to previous work
Survival | 12 months
  Success of the intervention, i.e no additional surgery during the study period due to lack of treatment effect or recurrence of symptoms.
Survival | 5 years
  Success of the intervention, i.e no additional surgery during the study period due to lack of treatment effect or recurrence of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Elin Swärd, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Department of hand surgery, Malmo university hospital, Malmo
  - Department of hand handsurgery, Södersjukhuset, Stockholm

REFERENCES:
- [Derived] Larsson SL, Tandrup T, Brogren E, Wilcke MK, Sward EM. Partial wrist denervation versus patient education and self-managed exercise therapy in patients with wrist osteoarthritis: study protocol for a randomized controlled trial. Trials. 2025 Oct 30;26(1):453. doi: 10.1186/s13063-025-09241-7. PMID 41168861